CLINICAL TRIAL: NCT03570957
Title: A Clinical Pharmacology Study of MT-2990 in Seasonal Allergic Rhinitis Patients (Single Dose Study)
Brief Title: A Clinical Pharmacology Study of MT-2990 in Seasonal Allergic Rhinitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-2990-J01
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MT-2990, Low dose (Experimental): Single intravenous dose
  Interventions: Drug: MT-2990; Drug: Placebo
- MT-2990, Low-middle dose (Experimental): Single intravenous dose
  Interventions: Drug: MT-2990; Drug: Placebo
- MT-2990, High-middle dose (Experimental): Single intravenous dose
  Interventions: Drug: MT-2990; Drug: Placebo
- MT-2990, High dose (Experimental): Single intravenous dose
  Interventions: Drug: MT-2990
- Placebo (Placebo Comparator): Single intravenous dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-2990 — MT-2990 solution for injection in vial
  Arms: MT-2990, High dose; MT-2990, High-middle dose; MT-2990, Low dose; MT-2990, Low-middle dose
Drug: Placebo — Placebo solution for injection in vial
  Arms: MT-2990, High-middle dose; MT-2990, Low dose; MT-2990, Low-middle dose; Placebo

SUMMARY:
The objective of this study is to investigate the safety, tolerability, and pharmacokinetics of MT-2990 in patients with Japanese cedar pollen-induced seasonal allergic rhinitis (JC-SAR). Additional objective of the study is to investigate the efficacy and pharmacodynamics profile of MT-2990 in an environmental exposure chamber (EEC) on Day 8, 29, 57, and 85.

ELIGIBILITY:
Inclusion Criteria:

* A body weight of 40 to 100 kg for female or 45 to 100 kg for male
* A body mass index of 18 to 30 kg/m2
* Subjects who have current history of JC-SAR in previous 2 consecutive years.
* Presence (CAP-RAST: ≥2) of IgE specific to Japanese cedar pollens and absence (CAP-RAST: ≤1) of IgE specific to other 4 allergens
* Presence of at least 2 symptoms, which are moderate to very severe, in 4 nasal symptoms (runny nose, sneezing, blocked nose, itchy nose) at any time point during allergen exposure in EEC at screening period

Exclusion Criteria:

* Presence of any symptoms of allergic rhinitis within 1 year except scattering season of cedar pollen or cypress pollen
* Subjects who have persistent symptom caused by allergen exposure in EEC at screening period until Day 1 (pre-dose)
* Underwent nasal surgery (include laser surgery) to improve nasal symptoms within 2 years
* Underwent specific immunotherapy or non-specific immunotherapy within 5 years
* Underwent medication of anti-histamine, oral mast cell stabilizer, leukotriene receptor antagonist, prostaglandin D2/thromboxane A2 receptor antagonist, Th2 cytokine inhibitor, corticosteroid (oral form, intra-nasal form, ocular form), or vasoconstrictor within 4 weeks
* Underwent medication of corticosteroid (injection form) or anti-IgE antibody within 6 months
* Subject who is concerned about exacerbation of the physical condition due to allergen exposure in EEC

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence of adverse events | Up to Day 113
Proportion of subjects who develop antibodies against MT-2990 in serum | Up to Day 113

SECONDARY OUTCOMES:
MT-2990 concentration in serum | Up to Day 113
Maximum observed serum concentration (Cmax) of MT-2990 | Up to Day 113
Measured time of maximum observed serum concentration (tmax) of MT-2990 | Up to Day 113
Apparent terminal elimination half-life (t1/2) of MT-2990 | Up to Day 113
AUC from time zero to the last measurable concentration (AUC0-last) of MT-2990 | Up to Day 113
AUC from time zero to infinity (AUC0-∞) of MT-2990 | Up to Day 113
Terminal elimination rate constant (kel) of MT-2990 | Up to Day 113
Apparent volume of distribution at steady state (Vss) of MT-2990 | Up to Day 113
Apparent volume of distribution during terminal phase after IV administration (Vz) of MT-2990 | Up to Day 113
Mean residence time from time zero to infinity (MRT0-∞) of MT-2990 | Up to Day 113
Apparent serum clearance (CL) of MT-2990 | Up to Day 113
Percentage of AUC obtained by extrapolation (%AUCex) of MT-2990 | Up to Day 113
Total nasal symptom score (TNSS) | Day 8, 29, 57, and 85
  Four nasal symptoms (runny nose, sneezing, blocked nose, and itchy nose) are recorded using a 5-point scale of 0 (none) to 4 (very severe). TNSS is sum of 4 nasal symptoms, score range is 0 to 16.
Total ocular symptom score (TOSS) | Day 8, 29, 57, and 85
  Two ocular symptoms (itchy eyes and watery eyes) are recorded using a 5-point scale of 0 (none) to 4 (very severe). TOSS is sum of 2 ocular symptoms, score range is 0 to 8.
Total symptom score (TSS) | Day 8, 29, 57, and 85
  TSS is TNSS plus TOSS.
Change from baseline in TNSS | Day 8, 29, 57, and 85
  Baseline is pre-exposure.
Change from baseline in TOSS | Day 8, 29, 57, and 85
Change from baseline in TSS | Day 8, 29, 57, and 85
Sum of TNSS during allergen exposure in EEC | Day 8, 29, 57, and 85
Sum of TOSS during allergen exposure in EEC | Day 8, 29, 57, and 85
Sum of TSS during allergen exposure in EEC | Day 8, 29, 57, and 85
AUC of TNSS after allergen exposure | Day 8, 29, 57, and 85
AUC of TOSS after allergen exposure | Day 8, 29, 57, and 85
AUC of TSS after allergen exposure | Day 8, 29, 57, and 85
Proportion of subjects with increased TNSS from baseline | Day 8, 29, 57, and 85
Proportion of subjects with increased TOSS from baseline | Day 8, 29, 57, and 85
Proportion of subjects with increased TSS from baseline | Day 8, 29, 57, and 85

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational Site, Tokyo, Japan